CLINICAL TRIAL: NCT00233168
Title: Promoting Adherence to TB Regimens in High Risk Youth
Brief Title: Effectiveness of Public Health Model of Latent Tuberculosis Infection Control for High-Risk Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Melbourne Hovell, Professor, Director/Center for Behavioral Epidemiology and Community Health, Graduate School of Public Health, San Diego State University, San Diego State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 323; R01HL068595 (NIH)
Record Dates: First submitted 2005-10-03; First posted 2005-10-05 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Lung Diseases; Tuberculosis
MeSH Terms: conditions — Lung Diseases; Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Peer medication adherence counseling
  Interventions: Behavioral: Adherence Program
- 2 (Active Comparator): Peer life skills counseling
  Interventions: Behavioral: Life Skills and Self-Esteem Training Program (Attention Control Arm)

INTERVENTIONS:
Behavioral: Adherence Program — 14 counseling sessions focusing on INH adherence conducted over 6 months, starting once per week and decreasing in frequency to once a month.
  Arms: 1
Behavioral: Life Skills and Self-Esteem Training Program (Attention Control Arm) — Peer counseling session covering life skills (e.g., communication skills, goal setting, self-esteem) training, 14 sessions over 6 months beginning once per week and decreasing in frequency over time to once per month.
  Arms: 2

SUMMARY:
This study will determine the differential cumulative mean number of isoniazid (INH) pills completed over 9 to 12 months for adolescents assigned to one of the following two groups: 1) peer adherence coaching, parent training, and self-esteem/life skills counseling; or 2) self-esteem/life skills counseling alone. The study will also estimate the costs and cost effectiveness of peer adherence coaching versus control procedures; this will be done from a provider and societal perspective.

DETAILED DESCRIPTION:
BACKGROUND:

Tuberculosis (TB) was responsible for almost one billion deaths in the 20th century. It is epidemic in the developing world and immigrants introduce TB to developed nations. TB control requires treatment for latent TB infection (LTBI) and active disease, as well as adherence to medical regimens. This study will determine the effectiveness of a public health model of LTBI control among high-risk adolescents. The integration of behavioral science, medical services, parent instruction, and assistance from schools and clinics (coordinated by the county health department) is based on recommendations from the Centers for Disease Control and Prevention (CDC). The effectiveness of this system is dependent, in part, on patient adherence.

DESIGN NARRATIVE:

The primary outcome of this study is adherence to an INH treatment regimen. For a given participant, adherence is assessed every 30 days, with the final outcome determined 12 months after treatment start date. Adherence is assessed using participant recall, urine testing for INH metabolites, pill counts, and medication event monitoring system (MEMS) caps.

The key secondary outcomes are parent knowledge and practice of intervention support procedures, parent knowledge of TB, self-esteem effects and life skills acquisition, cost and cost effectiveness of the intervention, and knowledge and practice of LTBI care by providers at participating community clinics.

ELIGIBILITY:
Inclusion Criteria:

* PPD positive
* San Diego County residents (without plans to relocate out of the county in the 12 months after study entry)
* Able to respond to the interview questions in English or Spanish
* Eligible for INH treatment

Exclusion Criteria:

* Receiving treatment in Mexico (due to differing medications and length of treatment)

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 263 (Actual)
Dates: Start 2003-09; Primary Completion 2007-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Number of INH pills taken | 12 months
  30-day recall of INH consumption measured monthly for up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Melbourne Hovell, Study Chair — San Diego State University
Locations (1):
- San Diego State University, San Diego, California, United States

REFERENCES:
- [Result] Hill LL, Hovell M, Blumberg E, Kelley N, Baird S, Sipan C, Schmitz K, Friedman L. Gaps between Adolescent Risk Behaviors and Disclosure during Outpatient Visits. Int J Family Med. 2013;2013:718568. doi: 10.1155/2013/718568. Epub 2013 Apr 24. PMID 23710357
- [Result] West JH, Blumberg EJ, Kelley NJ, Hill L, Sipan CL, Schmitz KE, Kolody B, Chambers CD, Friedman LS, Hovell MF. The Role of Parenting in Alcohol and Tobacco Use Among Latino Adolescents. J Child Adolesc Subst Abuse. 2013 Apr 1;22(2):120-132. doi: 10.1080/1067828X.2012.730359. Epub 2013 Feb 7. PMID 23439845
- [Result] West JH, Blumberg EJ, Kelley NJ, Hill L, Sipan CL, Schmitz KE, Ryan S, Clapp JD, Hovell MF. Does proximity to retailers influence alcohol and tobacco use among Latino adolescents? J Immigr Minor Health. 2010 Oct;12(5):626-33. doi: 10.1007/s10903-009-9303-2. PMID 19936923
- [Result] West JH, Blumberg EJ, Kelley NJ, Hill L, Sipan CL, Schmitz K, Kolody B, Madlensky L, Hovell MF. Latino parenting practices: a comparison of parent and child reports of parenting practices and the association with gateway drug use. J Ethn Subst Abuse. 2011;10(1):71-89. doi: 10.1080/15332640.2011.547800. PMID 21409705
- [Result] Hill L, Blumberg E, Sipan C, Schmitz K, West J, Kelley N, Hovell M. Multi-level barriers to LTBI treatment: a research note. J Immigr Minor Health. 2010 Aug;12(4):544-50. doi: 10.1007/s10903-008-9216-5. Epub 2008 Dec 16. PMID 19085104
- [Result] Schmitz KE, Hovell MF, Wong CA, Kelley NJ, Nilsen D, Blumberg EJ, Hill LL, Sipan CL, Kolody B, Chatfield DA. The reliability and practicality of the Arkansas method assay of isoniazid adherence. Clin Nurs Res. 2010 May;19(2):131-43. doi: 10.1177/1054773810363473. PMID 20435784
- [Derived] Hovell MF, Schmitz KE, Blumberg EJ, Hill L, Sipan C, Friedman L. Lessons learned from two interventions designed to increase adherence to LTBI treatment in Latino youth. Contemp Clin Trials Commun. 2018 Aug 16;12:129-136. doi: 10.1016/j.conctc.2018.08.002. eCollection 2018 Dec. PMID 30456327